CLINICAL TRIAL: NCT02474368
Title: Phase I Study Evaluating a Stereotactic Boost/Treatment for Recurrent or Metastatic Cancer of the Head and Neck
Brief Title: Study Evaluating a Stereotactic Boost/Treatment for Recurrent or Metastatic Cancer of the Head and Neck
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jonathan Schoenfeld, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-183
Record Dates: First submitted 2015-06-13; First posted 2015-06-17 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Head and Neck Carcinoma; Head and Neck Cancer Metastatic; Head or Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): * Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  * Cohort 1 (patients who have received prior radiation in the head and neck with gross unresectable disease)
    * Intensity Modulated Radiation Therapy (IMRT) : daily for 6 weeks
    * Cisplatin will be administered intravenously on predetermined days
    * Stereotactic Body Radiotherapy (SBRT)
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT); Drug: Cisplatin; Radiation: Stereotactic Body Radiotherapy (SBRT)
- Cohort 2 (Experimental): * Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  * Cohort 2 (patients with metastatic solid tumors of any histology who have targetable lesions within the head and neck) -- Stereotactic Body Radiotherapy (SBRT)
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy (IMRT)
  Arms: Cohort 1
Drug: Cisplatin
  Other Names: Platinol-AQ; Platinol
  Arms: Cohort 1
Radiation: Stereotactic Body Radiotherapy (SBRT)

SUMMARY:
This research study seeks to gain new knowledge about the addition of a carefully targeted "boost" dose of radiation as a possible treatment for recurrent or metastatic head or neck cancer. The name of the study intervention involved in this study is stereotactic body radiotherapy, which is a way of delivering radiation in a more precisely targeted way and with a higher dose than conventional radiotherapy.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

Stereotactic body radiation was developed as imaging and treatment capabilities on radiation treatment machines became more accurate and more precise. Like standard radiation therapy, stereotactic body radiation kills tumor cells by causing small breaks in the DNA of these cells. In this research study, the investigators are looking for the highest dose of the stereotactic radiation that can be given safely either alone, or as a 'boost dose' in combination with standard radiation and chemotherapy. Because stereotactic radiation is so precise, the investigators are testing whether it can be used to increase the dose to the primary tumor without significantly increasing the side effects; the goal is to improve the likelihood of killing the tumor and, in some cases, to complete the course of radiation in a shorter amount of time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* All cohorts:
* Participants must have a pathologic cancer diagnosis.
* No other active malignancy within the past 2 years, except for non-melanoma skin cancers or carcinoma in situ of the cervix.
* Only patients 18 years and older are eligible. There is no upper age limit but the patients must be able to medically tolerate the regimen. Adverse event data are currently unavailable on the use of SBRT for participants < 18 years of age, and thus children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (see Appendix A).
* Ability to understand and the willingness to sign a written informed consent document
* Cohort 1 (reirradiation in patients with head and neck cancers with gross unresectable disease):
* History of radiation to the head and neck area (defined as above the clavicles) greater than 6 months previous
* Pathologically proven recurrent disease or a second primary (squamous cell carcinoma of the head and neck, nasopharyngeal cancer, salivary gland cancer, or thyroid cancer) within the head and neck region, deemed to be unresectable or resected with gross residual disease remaining (determined by either operative/pathology report or post-surgical imaging)
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mcL (microliter)
  * Absolute neutrophil count > ↓1,500/mcL (microliter)
  * Platelets ≥100,000/mcL (microliter)
  * Total bilirubin within normal institutional limits
  * aspartate aminotransferase (AST (SGOT))/alanine aminotransferase (ALT (SGPT)) ≤ 2.5 x institutional upper limit of normal
  * Creatinine < 2 x upper limit of normal (ULN) or creatinine clearance ≥45 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
* Cohort 2 (patients with metastatic disease with targetable lesions within the head and neck):

  * Pathologically proven solid tumor (lymphomas excluded) with evidence of metastatic disease (including nodal disease)
  * Measurable disease within the head and neck region, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm and < 60 mm with neck CT scan. See section 10 for the evaluation of measurable disease.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* SBRT target size > 6 cm in maximum diameter (or greater than 100 cc in volume).
* Participants may not be receiving any other study agents.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because radiotherapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with SBRT, breastfeeding should be discontinued if the mother is treated with SBRT.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; or if diagnosed and treated within the past 2 years for cervical cancer in situ or basal cell or squamous cell carcinoma of the skin.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for interaction between conventional radiotherapy, SBRT and antiretroviral medications. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Patients who are planned to receive the following medications:

  * Granulocyte stimulating factor (G-CSF)
  * Bevacizumab
  * Cyclosporine
  * Anti-tumor necrosis factor agents
  * Amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2021-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of stereotactic body radiotherapy treatment (SBRT) when given as a boost in combination with cisplatin and intensity modulated radiation therapy (IMRT) | 1 Year
  Cohort 1: patients who have received prior radiation in the head and neck and currently have gross unresectable disease;
Maximum tolerated dose of stereotactic body radiotherapy treatment (SBRT) when given for disease metastatic to the head and neck | 1 year
  Cohort 2: Patients with metastatic disease with targetable lesions within the head and neck.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 1 Year
  Adverse events observed will be summarized in terms of type (organ affected or laboratory determination), severity (by National Cancer Institute, Common Toxicity Criteria for Adverse Effects - CTCAE v4 and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Local Control Rate | 1 Year
  Computed tomography (CT) and Positron emission tomography (PET) will be used to assess disease control within the field receiving radiation.
Regional Control Rate | 1 Year
  Computed tomography (CT) and Positron emission tomography (PET) will be used to assess disease control within the head and neck region.
Progression Free Survival using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 1 year
  Progression free survival will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol. The median progression free survival time will be estimated using standard life table methods.
Level of circulating activated T cells as an immune correlate of stereotactic treatment | 1 Year
  This will evaluate circulating immune cells before and after treatment and gene expression analysis focusing on delineating the immune components and immunologic milieu within the tumor before therapy.
Patient reported physical function before and after treatment | 1 year
  This will investigate changes in patient reported quality of life after treatment using the validated University of Washington Quality of Life Questionnaire (UW-QOL v4) composite score for physical function and comparing results obtained before and after treatment.
Patient reported social function before and after treatment | 1 year
  This will investigate changes in patient reported quality of life after treatment using the validated University of Washington Quality of Life Questionnaire (UW-QOL v4) composite score for social function and comparing results obtained before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Schoenfeld, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No